CLINICAL TRIAL: NCT02913547
Title: Safety, Efficacy and Usage Compliance of the Silk'n HST Home Use Device for Treating Periorbital Wrinkles and Improving Skin Appearance
Brief Title: Silk'n HST for Wrinkle Reduction - Clinical Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO109828
Record Dates: First submitted 2016-09-11; First posted 2016-09-23 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2016-09

CONDITIONS: Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Each subject will serve as his/her own control, while comparing results before treatment, and after 6 weeks of treatment.
  Intervention includes treatment with the Silk'n HST on the periorbital areas as instructed in the user's manual.
  Interventions: Device: Silk'n HST

INTERVENTIONS:
Device: Silk'n HST — Treatment with Silk'n HST on the periorbital area as instructed in the user's manual

SUMMARY:
The objective of the study is to evaluate the safety, efficacy and usage compliance of the home-use device Silk'n HST for self-treatment of periorbital wrinkles and skin laxity and improvement of skin appearance.

DETAILED DESCRIPTION:
This is a single arm prospective study of 18 weeks aimed to evaluate the safety and efficiency of Silk'n HST treatment on the periorbital areas. 30 subjects will be enrolled by a single USA clinical site. Throughout the trial there will be 3 pre-scheduled face to face treatment visits, as well as additional 18 independent treatments at home. 2 additional follow-up visits will be conducted 1 and 3 months following treatment end. In addition, 2 maintenance treatment will be conducted independently at home once a month following treatment end.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 35-65.
2. The subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side effects, and sign the Informed Consent Form, including the permission to use photography (forms attached).
3. The subjects should be willing to comply with the study procedure and schedule, including the follow up visits, and will refrain from using any other or similar treatment technologies (i.e., Laser, RF, IR) for the facial condition.
4. The subjects will carry on with their usual diet and exercise and will not have a significant weight change during the study.
5. The subject is able to read the User Manual in English.
6. Subjects should have II-VI Fitzpatrick wrinkle score as indicated on the Fitzpatrick Wrinkle and Elastosis Scale (see Table 1).
7. Negative results in a urine pregnancy test.

Exclusion Criteria:

1. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
2. Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance.
3. Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles per investigator's discretion.
4. Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases per investigator's discretion.
5. Pregnancy or nursing, as well as 3-6 months post-childbirth.
6. History of bleeding coagulopathies, or prolonged use of anticoagulants (daily aspirin dosing of 81 mg is acceptable).
7. Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medication per investigator's discretion.
8. Subjects with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regime.
9. Poorly controlled endocrine disorders, such as diabetes or thyroid abnormality per investigator's discretion.
10. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash per investigator's discretion.
11. History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin per investigator's discretion.
12. Any surgery in treated area within 3 months prior to treatment or before complete healing.
13. Injected fillers in the last 6 months and Botox in the last week.
14. Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
15. As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the subject.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
reduction of wrinkle severity according to the Fitzpatrick wrinkle scale | 18 weeks
  measurements were accomplished via standardized photographs blinded evaluation.

SECONDARY OUTCOMES:
subjective wrinkle improvement as measured by satisfactory questionnaires | 18 weeks
  A subjective impression of improvement in wrinkle appearance following 6 weeks treatment, 3 months following treatment end.

IPD SHARING:
Plan to Share IPD: Undecided